CLINICAL TRIAL: NCT05248516
Title: Simplified Treatment of Children With Low WAZ in Mali. A Randomized Controlled Trial
Brief Title: ComPAS Low-WAZ RCT Mali
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Rescue Committee (Other)
Collaborators: University of the Sciences, Techniques and Technologies of Bamako (Other); Ministry of health, Mali (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H 1.00.033
Record Dates: First submitted 2022-01-27; First posted 2022-02-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Acute Malnutrition in Infancy; Acute Malnutrition in Childhood; Underweight
Keywords: wasting; stunting; underweight; malnutrition; ready-to-use therapeutic food; acute malnutrition; randomized controlled trial; weight-for-age z-score; mid-upper-arm circumference; Mali
MeSH Terms: conditions — Thinness; Cachexia; Growth Disorders; Malnutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): no nutritional treatment administered
  Interventions: Dietary Supplement: No nutritional treatment
- Simplified treatment (Experimental): children are provided with 1 sachet of RUTF until discharge
  Interventions: Dietary Supplement: Simplified dose of ready-to-use therapeutic food (RUTF)
- Standard treatment (Active Comparator): children are provided nutritional treatment according to their weight-for-height z-score (WHZ) and their weight:
  1. children with a WHZ<-3 will receive 200kcal/kg/d of nutritional product until discharge
  2. children with a WHZ between -3 and -2 are provided with 1 sachet of RUTF until discharge
  3. children with a WHZ >= -2 will not be provided any nutritional treatment
  Interventions: Dietary Supplement: Standard dose of ready-to-use therapeutic food (RUTF)

INTERVENTIONS:
Dietary Supplement: Simplified dose of ready-to-use therapeutic food (RUTF) — In the simplified arm all children receive the same dose: 1 sachet of RUTF/day. This until discharge from treatment.
  Recovery from treatment will be defined as WAZ>= -3 on 2 consecutive visits. A maximum of 12 treatment weeks are allowed before declaring non-response. Defaulting will be declared after 2 consecutively missed visits.
  Arms: Simplified treatment
Dietary Supplement: Standard dose of ready-to-use therapeutic food (RUTF) — In the standard arm, children will receive different doses of RUTF depending on their WHZ category and weight.
  1. children with a WHZ<-3 will receive the equivalent of 200kcal/kg/d of RUTF until discharge.
  2. children with a WHZ between -3 and -2 will receive 1 sachet (500kcal) of RUTF per day until discharge.
  3. children with a WHZ>=-2 will receive no nutritional treatment.
  Recovery from treatment will be defined as WHZ>= -2 on 2 consecutive visits. A maximum of 12 treatment weeks are allowed before declaring non-response. Defaulting will be declared after 2 consecutively missed visits.
  Arms: Standard treatment
Dietary Supplement: No nutritional treatment — no nutritional treatment will be provided to children in the control arm.
  Arms: Control

SUMMARY:
Admissions criteria which treat children with only low mid-upper arm circumference (MUAC) or children with low weight-for-height z-score (WHZ) are not aligned with the evidence on which children are at risk of mortality. An analysis of community-based cohort data from Senegal found that a combination of weight-for-age z-score (WAZ) and MUAC criteria identified all children at risk of near-term death associated with severe anthropometric deficits. This finding has led to the suggestion that WAZ<-3 could be added as an independent admissions criterion for therapeutic feeding programs currently admitting children with MUAC<125 mm. However, there is little evidence to inform the debate about whether children with MUAC ≥125 mm and WAZ<-3 would benefit from treatment and, if so, what treatment protocol should be used.

This study will address whether children with WAZ <-3 but MUAC ≥125 mm benefit from therapeutic feeding and whether a simplified protocol is at least as effective as the more complicated weight-based standard protocol for this population.

The study will be a prospective, multi-center, individually randomized controlled trial (RCT). Children aged 6-59 months presenting with MUAC ≥125 mm and WAZ<-3 will be randomized to one of three study arms.

The primary objective of this study is to assess whether therapeutic feeding with a simplified protocol (1 sachet RUTF/day) results in superior nutritional outcomes compared to no therapeutic feeding AND non-inferior nutritional outcomes compared to the WHZ and weight based dosing regimen currently used in CMAM treatment 2 months after diagnosis among children aged 6-59 months with MUAC ≥125 mm and WAZ<-3 .

The primary outcome is the mean WAZ of children. Secondary outcomes include a) proportion of children with WAZ <-3, b) mean MUAC of children, c) proportion of children with MUAC < 125 mm, d) mean WHZ, mean HAZ, e) proportion of children with WHZ<-3 or HAZ<-3, f) change in WAZ, MUAC, WHZ, HAZ from enrolment to endpoint g) mean skinfold thickness measure.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 and 59 months
* MUAC ≥125 mm
* WAZ <-3
* Living in the study catchment area
* Expects to be able to continue follow-up visits for next 6 months

Exclusion Criteria:

* nutritional edema
* Known peanut or milk allergy
* Severe illnesses requiring inpatient level treatment (according to IMCI guidelines)
* Medical condition affecting food intake (lip and palate cleft, handicap etc.)
* Has already taken part in the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
weight-for-age z-score (WAZ) | 2 months after enrolment
  the primary outcome is a continuous outcome: a higher WAZ indicates of a positive outcome. To construct WAZ at any point in time, children's age will be calculated based on their age at admission and their weight will be measured at each time point with 0.1kg precision. WAZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.

SECONDARY OUTCOMES:
weight-for-age z-score (WAZ) | 6 months after enrolment
  the secondary outcome is a continuous outcome: a higher WAZ indicates a positive outcome. To construct WAZ at any point in time, children's age will be calculated based on their age at admission and their weight will be measured at each time point with 0.1kg precision. WAZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
weight-for-age z-score (WAZ) <-3 | both at 2 and 6 months post-enrolment
  this outcome is binary: a higher proportion of WAZ<-3 indicates a negative outcome. To construct WAZ at any point in time, children's age will be calculated based on their age at admission and their weight will be measured at each time point with 0.1kg precision. WAZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
weight-for-height z-score (WHZ) | both at 2 and 6 months post-enrolment
  this outcome is a continuous outcome: a higher WHZ indicates a positive outcome. To construct WHZ at any point in time, children's height and weight will be measured at each time point: height with 0.1cm precision and weight with 0.1kg precision. WHZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
weight-for-height z-score (WHZ) <-3 | both at 2 and 6 months post-enrolment
  this outcome is binary: a higher proportion of WHZ<-3 indicates a negative outcome. To construct WHZ at any point in time, children's height and weight will be measured at each time point: height with 0.1cm precision and weight with 0.1kg precision. WHZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
height-for-age z-score (HAZ) | both at 2 and 6 months post-enrolment
  this outcome is a continuous outcome: a higher HAZ indicates a positive outcome. To construct HAZ at any point in time, children's age will be calculated based on their age at admission and their height will be measured at each time point with 0.1cm precision. HAZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
height-for-age z-score (HAZ) <-3 | both at 2 and 6 months post-enrolment
  this outcome is binary: a higher proportion of HAZ<-3 indicates a negative outcome. To construct HAZ at any point in time, children's age will be calculated based on their age at admission and their height will be measured at each time point with 0.1cm precision. HAZ will be calculated using zscore06 fonction in STATA that is based on the WHO growth reference data specific to each gender.
Mid-upper-arm circumference (MUAC) | both at 2 and 6 months post-enrolment
  this outcome is a continuous outcome: a higher MUAC indicates a positive outcome. MUAC will be measured using a while MUAC tape with a precision of 1mm.

OTHER OUTCOMES:
subscapular skin-fold thickness in millimeters | 2 and 6 months post-enrolment
  this outcome is a continuous outcome. there are currently no internationally accepted standards for the skinfold measure of young children. we will thus report the mean and any other relevant data on this and discuss the results in light of past research.
proportion having developed a mid-upper-arm circumference <125mm | 6 months post-enrolment
  the proportion of children that exit the study with a MUAC<125mm at any point in time will be estimated. MUAC will be measured at each visit using a while MUAC tape with a precision of 1mm.
tricep skin-fold thickness in millimeters | 2 and 6 months post-enrolment
  this outcome is a continuous outcome. there are currently no internationally accepted standards for the skinfold measure of young children. we will thus report the mean and any other relevant data on this and discuss the results in light of past research.
fat-free mass in kg | 2 and 6 months post-enrolment
  this outcome is a continuous outcome obtained through bioelectrical impedance analysis and applying a suitable equation to obtain fat-free mass estimations from weight and impedance.
fat mass in kg | 2 and 6 months post-enrolment
  this outcome is a continuous outcome obtained through bioelectrical impedance analysis and applying a suitable equation to first obtain fat-free mass estimations from weight and impedance and then by substracting fat-free mass from weight.
fat-free mass index in kg/m2 | 2 and 6 months post-enrolment
  this outcome is a continuous outcome obtained through bioelectrical impedance analysis and applying a suitable equation to obtain fat-free mass estimations from weight and impedance and indexing fat-free mass to height squared to adjust for differences in size.
fat mass index in kg/m2 | 2 and 6 months post-enrolment
  this outcome is a continuous outcome obtained through bioelectrical impedance analysis and applying a suitable equation to first obtain fat-free mass estimations from impedance and weight and then substracting fat-free mass from weight and indexing the obtained fat mass to height squared to adjust for differences in size.
hemoglobin (g/l) | 2 and 6 months
  this is a continuous outcome and will be obtained through HemoCue measurement of peripheral blood
anaemia | 2 and 6 months
  this is a binary outcome and will be obtained through hemoglobin measurement of peripheral blood and categorising Hb<11g/l as anaemic.

CONTACTS AND LOCATIONS:
Locations (11):
- Mali (11):
  - Dilly, Nara, Koulikoro
  - Gassambarou, Nara, Koulikoro
  - Goumbou, Nara, Koulikoro
  - Kaloumba, Nara, Koulikoro
  - Karfabougou, Nara, Koulikoro
  - Koira, Nara, Koulikoro
  - Koronga, Nara, Koulikoro
  - Madina-Kagoro, Nara, Koulikoro
  - Nara Central, Nara, Koulikoro
  - Sampaga, Nara, Koulikoro
  - Tiapato, Nara, Koulikoro

IPD SHARING:
Plan to Share IPD: Yes
The investigators are planning on making data underlying publications available through on-line data repositories such as Zenodo. This data would be de-identified prior to sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP and ICF will be published with the main results. The SAP will also be made available through clinicaltrials.gov prior to trial data collection completion. The study data underlying the key findings will be made freely available once analysis is complete and results published for the primary and secondary objectives and outcomes.
Access Criteria: Study protocol, SAP and ICF will be openly available via the publication. The study data will be made freely available from Zenodo or similar data repository.

REFERENCES:
- [Derived] Kangas ST, Ouedraogo CT, Tounkara M, Ouoluoguem B, Coulibaly IN, Haidara A, Diarra NH, Diassana K, Tausanovitch Z, Ritz C, Wells JC, Briend A, Myatt M, Radin E, Bailey J. Nutritional treatment of children 6-59 months with severely low weight-for-age z-score: a study protocol for a 3-arm randomized controlled trial. Trials. 2024 Jan 8;25(1):30. doi: 10.1186/s13063-023-07890-0. PMID 38191436